CLINICAL TRIAL: NCT05450159
Title: Evaluating the Acceptability and Feasibility of an Evidence-based and User-informed Approach to Refreshing Older Adults' Driving Skills (ROADSkills)
Brief Title: The Refreshing Older Adults' Driving Skills (ROADSkills) Program
Acronym: ROADSkills
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: Ontario Ministry of Transportation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14707
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Drive

STUDY DESIGN:
Intervention Model Description: 2-arm, parallel-group, double-blinded Randomized Controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Video recordings of the on-road evaluation wil be scored by an independent (outcomes) assessor blinded to participant identity, group allocation, and whether the drive was from the baseline or after the intervention. Blinding will be enforced by randomly assigning a unique number to each video after a participant has completed their 3 months of driver monitoring. Videos will be forwarded to the rater in batches of 8-10.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will watch their respective training video individually approximately four to six weeks after their baseline visit. Each training video will be 20-25 minutes in length where they will receive voice-over feedback on their driving from a member of the study team alongside video clips taken from the device of their behind-the-wheel performance. They will also receive a written summary of their feedback to keep at the end of their feedback session.
  Interventions: Behavioral: ROADskills program
- Control group (Active Comparator): Four to six weeks after their first baseline visit, control group participants individually will watch a 30-minute (generic) video that describes the benefits and challenges of aging-in-place that discusses the importance of community mobility in later life. At the end of their session, participants will be given a government brochure on this topic.
  Interventions: Behavioral: Healthy Aging

INTERVENTIONS:
Behavioral: ROADskills program — Participants in the intervention arm of the study will watch a 30-minute personalized video on their driving that uses information compiled from a GPS device that will be installed in their vehicle during their baseline visit.
  Arms: Intervention group
Behavioral: Healthy Aging — Participants in active comparator arm of the study will watch a 30-min video and receive a written brochure that provide tips for maintaining a healthy lifestyle in later life, including the importance of community mobility.
  Arms: Control group

SUMMARY:
Drivers aged 65+ depend on their car(s) to get to the places and see the people that are important to them. Losing a license in later life has been linked to higher rates of loneliness, depression, and even admission to long-term care; a fact that is particularly relevant when considering the impact of the COVID-19 pandemic. While drivers in this age group are among the safest on the road, they have one of the highest risks of collision when distance driven is considered and are more likely to be seriously injured or killed. Motor vehicle crashes and falls are the top causes of injury-related hospitalizations in seniors. Through a partnership with older adults, driving instructors, and health professionals, we developed the Refreshing Older Adult Driving Skills (ROADSkills) program. This program uses a Global Positioning System (GPS) device that can be placed in people's cars, which can track their real-world, everyday driving patterns, including speeding and hard braking, alongside video data of their behind-the-wheel behaviour. Using this data, a personalized video will be created using information captured by the device in the older driver's car. This study will determine if the older drivers who receive this video feedback perform better than those who do not receive such feedback. Because this is the first time a study will use this type of behavioural intervention, we are interested in hearing from older drivers about their experience of participating in the study. The findings will help us to design a larger, national study of the ROADSkills program in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65-79 to reduce co-intervention bias, as the Ministry of Transportation has a Senior Driver Renewal program that screens drivers aged 80 and older
* Hold a valid driver's license
* Owner and access to insured vehicle
* Speak and understand English fluently
* Visited an optometrist in last two years
* if corrective lens are required for driving, prescriptions should be up-to-date

Exclusion Criteria:

* If participated in a recent Randomized Controlled Trial that examined the effectiveness of video-based intervention, will be excluded due to potential for bias
* Known serious or terminal illness or presence of contraindications for driving
* Performance on cognitive screening: 1) score of < 21 on the Montreal Cognitive Assessment (MoCA; Nasreddine et al., 2005) 2) taking longer than 180 seconds or 3 or more errors on the Trail Making Test B (Bowie & Harvey, 2006).

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
weighted electronic Driving Observation Schedule (eDOS) | 3 months
  The weighted eDOS (Chen et al., 2020; Mazer et al., 2021) will be used to evaluate the behind-the-wheel performance of older drivers. The weighted eDOS accounts for route complexity where a total score is calculated, as the sum of errors weighted for its risk level. For each driving error, a weight is given (1=low risk; 2=moderate risk; 3=high risk) based on the type of error and the environment where it was made. For example, no signal at intersection with only one lane in low speed is considered a low-risk error whereas an inappropriate gap when making a left turn across more than one lane of traffic is a high-risk error. The weighted eDOS will be scored by a trained rater (blinded) using the GPS data of a 20-25- minute route. The weighted eDOS emerged from research examining the real-world driving of older drivers and has good inter-rater reliability, internal consistency and ecological validity; acceptability among older drivers was high (Koppel et al., 2016; 2017).

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster Automotive Resource Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen YT, Gelinas I, Mazer B. Development of a weighted scoring system for the Electronic Driving Observation Schedule (eDOS). MethodsX. 2020 Oct 12;7:101099. doi: 10.1016/j.mex.2020.101099. eCollection 2020. PMID 33224736
- [Background] Mazer B, Chen YT, Vrkljan B, Marshall SC, Charlton JL, Koppel S, Gelinas I. Comparison of older and middle-aged drivers' driving performance in a naturalistic setting. Accid Anal Prev. 2021 Oct;161:106343. doi: 10.1016/j.aap.2021.106343. Epub 2021 Aug 18. PMID 34418687
- [Background] Koppel S, Charlton JL, Langford J, Di Stefano M, MacDonald W, Vlahodimitrakou Z, Mazer BL, Gelinas I, Vrkljan B, Eliasz K, Myers A, Tuokko HA, Marshall SC. Driving Task: How Older Drivers' On-Road Driving Performance Relates to Abilities, Perceptions, and Restrictions. Can J Aging. 2016 Jun;35 Suppl 1:15-31. doi: 10.1017/S0714980816000015. Epub 2016 Mar 29. PMID 27021591
- [Background] Koppel S, Charlton JL, Richter N, Di Stefano M, Macdonald W, Darzins P, Newstead SV, D'Elia A, Mazer B, Gelinas I, Vrkljan B, Eliasz K, Myers A, Marshall S. Are older drivers' on-road driving error rates related to functional performance and/or self-reported driving experiences? Accid Anal Prev. 2017 Jun;103:1-9. doi: 10.1016/j.aap.2017.03.006. Epub 2017 Mar 31. No abstract available. PMID 28365398